CLINICAL TRIAL: NCT07222865
Title: Towards Realtime High-resolution Treatment Monitoring in Humans: Using Ultrasound Imaging to Monitor Low-intensity Focused Ultrasound Neuromodulation
Brief Title: tFUS Imaging & LIFU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study does not need to be registered. Study team wishes to withdraw registration
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 25-953
Record Dates: First submitted 2025-10-01; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Brain Imaging

STUDY DESIGN:
Intervention Model Description: All participants will complete all study visits - fMRI + tasks, tFUS + tasks, and tFUS + LIFU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Arm 1 - all participants (Experimental): All participants will receive two imaging modalities with corresponding tasks to compare imaging modalities.
  Interventions: Device: Feasibility of imaging using tFUS

INTERVENTIONS:
Device: Feasibility of imaging using tFUS — Imaging using transcranial functional ultrasound.

SUMMARY:
This study is investigating a new method of brain imaging - transcranial functional ultrasound (tFUS). We are comparing the imaging capabilities with functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
A battery of tasks will be performed under two imaging conditions. Magnetic Resonance Imaging and transcranial functional ultrasound imaging. Tasks include a breath hold task, an e-stim task, and low-intensity focused ultrasound neuromod.

ELIGIBILITY:
Inclusion Criteria:

* See above.

Exclusion Criteria:

* Claustrophobia
* Contraindications to MRI (neurostims, metal implants, pacemakers, etc)
* Contraindications to CT (pregnancy)
* Active medical disorders with CNS effects (e.g. Alzheimers)
* History of neurological disorder
* History of head injury with LOC > 10 min
* History of alcohol or drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Detecting task-evoked changes | The duration of each task - ~10 minutes.
  Detecting task-evoked changes using tFUS imaging

SECONDARY OUTCOMES:
Detecting LIFU induced neural activity | During LIFU application, ~2 min.
  Detection in changes of neural activity during LIFU using tFUS

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No